CLINICAL TRIAL: NCT03183661
Title: Follow-up Study to Evaluate the Safety of ALLO-ASC-CD in the Subjects With Crohn´s Disease(ALLO-ASC-CD-101)
Brief Title: A Follow-up Study to Evaluate the Safety of ALLO-ASC-CD in ALLO-ASC-CD-101 Clinical Trial
Status: Recruiting | Type: Observational
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-ASC-CD-102
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALLO-ASC-CD injection: Subjects with ALLO-ASC-CD injection in phase 1 clinical trial of ALLOASC-CD-101
  Interventions: Biological: ALLO-ASC-CD

INTERVENTIONS:
Biological: ALLO-ASC-CD — ALLO-ASC-CD is intravenous infusion containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells are directed to injured tissue, and reduce inflammation. Furthermore their immunomodulatory effects are significant for treating immune-related disease. Finally, ALLO-ASC-CD may provide a new option in treating a crohn's disease. This study is a follow-up study without intervention.
  Other Names: Allogenic adipose-derived mesenchymal stem cell

SUMMARY:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-CD injection in phase 1 clinical trial (ALLO-ASC-CD-101) for 36 months.

DETAILED DESCRIPTION:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-CD injection in phase 1 clinical trial (ALLO-ASC-CD-101) for 36 months.

ALLO-ASC-CD is intravenous infusion containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells are directed to injured tissue, and reduce inflammation. Furthermore their immunomodulatory effects are significant for treating immune-related disease, such as crohn's disease. Finally, ALLO-ASC-CD may provide a new option in treating a crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are injected with ALLO-ASC-CD in phase 1 clinical trial of ALLO-ASC-CD-101.
2. Subjects who are able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Subjects who are considered not suitable for the study by the principal investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject is enrolled who are injected ALLO-ASC-CD intravenous infusion in phase 1 clinical trial of ALLO-ASC-CD-101.
Sampling Method: Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2016-11-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 36 months
  Evaluation of AE

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hee Cheon, Ph D, Principal Investigator — Yonsei University; Joo Sung Kim, Ph D, Principal Investigator — Seoul National University Hospital; Young Ho Kim, Ph D, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided